CLINICAL TRIAL: NCT01280149
Title: Reduction of IgE Antibody in Human Allergic Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Paul Greenberger, Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BB-IND 4458
Record Dates: First submitted 2011-01-18; First posted 2011-01-20 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: substance P; allergic rhinitis; allergen immunotherapy
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis, Allergic | interventions — Substance P

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- substance P-low dose allergen (Experimental): Substance P injections with 8 sequential, increasing doses of allergen
  Interventions: Biological: substance P; Biological: substance P injections
- substance P-moderate dose allergen (Experimental): Substance P with sequential, increasing doses of allergen
  Interventions: Biological: substance P; Biological: substance P injections
- substance P-low/moderate dose allergen (Experimental): substance P with 16 sequential increasing doses of allergen
  Interventions: Biological: substance P; Biological: substance P injections
- substance P-placebo (Active Comparator): Placebo injections of substance P and placebo
  Interventions: Biological: substance P; Biological: substance P injections
- placebo-low dose allergen (Experimental): Placebo injections with 8 sequential increasing low dose allergen injections
  Interventions: Biological: substance P; Biological: substance P injections
- placebo-placebo (Placebo Comparator): substance P placebo and allergen placebo (weekly)
  Interventions: Biological: substance P; Biological: substance P injections

INTERVENTIONS:
Biological: substance P — injections of substance P and low dose allergen or placebo
Biological: substance P injections — injections of substance P for 8 weeks

SUMMARY:
The purpose of this study is to determine whether a neuropeptide, substance P, when injected along with an allergen, such as ragweed, can reduce allergic reactivity.

DETAILED DESCRIPTION:
Allergic Rhinitis (Hay fever) affects many children and adults and is a risk factor for development of asthma. This study utilizes the neurotransmitter, substance P, a small molecule which is present in nerve endings, the brain, skin, lungs and the gastrointestinal tract. Subjects will receive substance P and a low dosage of an allergen, such as ragweed in an attempt to reduce allergic reactivity.

ELIGIBILITY:
Inclusion Criteria:

* positive immediate type skin test to ragweed or grass pollen or a third (standardized) allergen if both ragweed and grass pollen allergen are not positive
* volunteers should be available for allergen injections and then cutaneous titrations for approximately 1 year from the start of the enrollment period

Exclusion Criteria:

* volunteer is pregnant or lactating
* abnormal electrocardiogram for subjects over 50 years of age
* use of beta adrenergic antagonists or tricyclic antidepressants

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2017-06-20 (Actual); Study Completion 2017-06-20 (Actual)

PRIMARY OUTCOMES:
CBER ID50 skin test result | 1 to 6 months after completing injections
  The ID50 skin test result utilizes FDA CBER methodology to determine the change in allergic skin reactivity to ragweed and grass pollen allergens.

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Greenberger, M.D., Principal Investigator — Northwestern University Feinberg School of Medicine
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No